CLINICAL TRIAL: NCT05926336
Title: To Compare the Effects of Intraoperative Use of Intravenous Anesthetics Propofol and Inhaled Anesthetics Sevoflurane on the Prognosis of Patients Undergoing Surgery for Primary Brain, Liver, Lung, and Ovarian Cancer Tumors and the Investigation of Its Mechanism of Action
Brief Title: The Effects of Using Different Anesthetics on the Prognosis of Primary Tumors and Its Mechanism of Action
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20230075
Record Dates: First submitted 2023-05-26; First posted 2023-07-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer; Brain Tumor; Liver Cancer; Ovarian Cancer
Keywords: Propofol; Sevoflurane; Survival
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms; Liver Neoplasms; Ovarian Neoplasms | interventions — Propofol; Sevoflurane; Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Experimental): The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3).
  Interventions: Drug: Sevoflurane
- Propofol (Experimental): The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Other Names: total intravenous anesthesia
  Arms: Propofol
Drug: Sevoflurane — The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3 MAC)
  Other Names: inhalation anesthesia
  Arms: Sevoflurane

SUMMARY:
1. Eligible participants were assessed prior to anesthesia. After the patient is admitted to the hospital, the subject's consent form is explained, and the consent form must be signed before the operation.
2. This is a two-arm, parallel-group randomized clinical trial.In the preoperative waiting area, the patients are randomly assigned and divided into two groups according to the allocation sequence table (corresponding to 1:1 randomization) generated by the computer. The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system. The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3). During the operation, the dose of anesthetic drugs (propofol/fentanyl /remifentanil and sevoflurane/cisatracurium/rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value and Entropy (or BIS) value at 40-60in both groups. The following patient data were recorded, the type of anesthesia, sex, age at the time of surgery, preoperative Karnofsky performance status (KPS) score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), ASA physical status scores, tumor marker ,tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/fentanyl) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, 3-year and 5-year overall survival and Karnofsky performance status score were recorded.

DETAILED DESCRIPTION:
During the operation, the dose of anesthetic drugs (propofol/ fentanyl /remifentanil and sevoflurane/ cisatracurium/ rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value and Entropy (or BIS) value at 40-60in both groups. The following patient data were recorded, the type of anesthesia, age at the time of surgery, preoperative Karnofsky performance status (KPS) score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), ASA physical status scoress, tumor marker , tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/ fentanyl/ propofol) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, and 3-year overall survival and Karnofsky performance status score were recorded.

ELIGIBILITY:
Inclusion Criteria:

* eighteen to eighty-year-old
* ASA class I-III patients
* Elective surgery for brain, liver, lungs, ovarian cancer under general anesthesia

Exclusion Criteria:

* Severe mental disorder, poor liver function, pregnant or lactating women, morbidly obese, allergy to any of the drugs used in this study, recurrent tumor or repeat surgery, biopsy cases, incomplete outcome-data, palliative treatment after surgery, simultaneous treatment of other malignancies, emergency surgery, presence of other malignant tumors, combined propofol and inhalation anesthesia or other anesthetics, such as ketamine or dexmedetomidine, diagnosed as benign brain, liver, lungs, ovarian cancer、cell carcinoma or other metastatic.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1316 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  6-month overall survival, 1-year overall survival, and 3-year overall survival
The presence of disease progression | From the date of surgery until the date of first documented progression (recurrence or metastasis),assessed up to 36 months
  From the date of surgery until the date of first documented progression (recurrence or metastasis) or date of death from any cause, assessed up to 36 months

SECONDARY OUTCOMES:
Postoperative complications | The period from the day of surgery to postoperative 30 days
  Clavien-Dindo classification, and other postoperative complications
Karnofsky performance status score | postoperation 6 months, postoperation 12 months,postoperation 36 months.
  Karnofsky performance score, from 100 to 0, where 100 is perfect health and 0 is death. The lower the Karnofsky performance score, the worse the likelihood of survival.
Length of hospital stays | from the day of surgery to dischage, assessed up to 30 days
  the length of stays in general ward and ICU

OTHER OUTCOMES:
time of operation and anesthesia | from start to end of the procedure
  record the time the opeartion and anesthesia
blood loss | from start to end of the procedure
  record the blood loss (ml)
volume of blood transfusion | from start to end of the procedure
  volume of blood transfusion (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Fu Wu, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan